CLINICAL TRIAL: NCT00978185
Title: The Effectiveness and Cost Effectiveness of Acupressure for the Control and Management of Chemotherapy-related Nausea.
Brief Title: Acupressure Wristbands or Standard Care in Controlling Nausea Caused by Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manchester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Supportive Care
Other Study IDs: CDR0000649812; UM-ACMCN; EU-20971
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-09

CONDITIONS: Anxiety Disorder; Nausea and Vomiting; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: nausea and vomiting; anxiety disorder; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Anxiety Disorders; Nausea; Vomiting | interventions — Acupressure

INTERVENTIONS:
Other: medical chart review
Other: questionnaire administration
Procedure: acupressure therapy
Procedure: quality-of-life assessment
Procedure: sham intervention
Procedure: standard follow-up care

SUMMARY:
RATIONALE: Acupressure wristbands may prevent or reduce nausea caused by chemotherapy. It is not yet known whether acupressure wristbands are more effective than standard care in controlling acute and delayed nausea.

PURPOSE: This randomized phase III trial is studying acupressure wristbands to see how well they work compared with standard care in controlling nausea caused by chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To assess the clinical effectiveness of self-acupressure using wristbands in addition to standard care in the management of chemotherapy-induced (acute and delayed) nausea compared to patients receiving standard care with sham-acupressure wristbands and standard care alone.

Secondary

* To assess the cost effectiveness and extent of use of usual care in patients using acupressure wristbands in addition to standard care for the management of chemotherapy-induced nausea compared to patients receiving standard care with sham-acupressure wristbands and standard care alone.
* To assess the level of quality of life in patients using acupressure and standard care alone.
* To assess the clinical effectiveness of self-acupressure using wristbands in addition to standard care in the management of chemotherapy-induced (acute and delayed) vomiting compared to patients receiving standard care with sham-acupressure wristbands and standard care alone.
* To ascertain for which emetogenic level of chemotherapy regimens (i.e., high, moderate, or low emetogenic chemotherapy) self-acupressure using wristbands in addition to standard care is more or less effective in terms of nausea compared to patients receiving standard care with sham-acupressure wristbands and standard care alone.
* To ascertain whether any improvement in chemotherapy-induced nausea and vomiting from using acupressure wristbands is different in males and females.
* To ascertain whether there is an age effect from the use of acupressure wristbands in relation to chemotherapy-induced nausea and vomiting.

OUTLINE: Patients are stratified according to gender, age in years (16 to 24 vs >24 to 50 vs > 50), and level of emetogenic chemotherapy (high vs moderate vs low). Patients are randomized to 1 of 3 intervention arms:

* Arm I (acupressure group): Patients receive standard antiemetics comprising an oral 5-HT3 receptor antagonist (i.e., Zofran) and oral or IV dexamethasone before and for 3 days post-chemotherapy (for highly emetic chemotherapy); an oral 5-HT3 receptor antagonist (i.e., Zofran) and dexamethasone IV before chemotherapy and a 5-HT3 receptor antagonist or dexamethasone for 2 days post-chemotherapy (for moderately emetogenic chemotherapy); or oral dexamethasone before chemotherapy (for low-emetogenic chemotherapy). Beginning on the morning before chemotherapy, patients wear a pair of SeaBand™ elastic wristbands on each arm for 7 days. Each wristband has a 1-cm protruding round plastic button (stud) pressing the P6 acupoint, located on the anterior surface of the forearm, approximately three-finger width up from the crease of the wrist between the tendons of the Palmaris longus and flexor carpi radialis.
* Arm II (sham acupressure group): Patients receive standard antiemetics as in arm I. Beginning on the morning before chemotherapy, patients wear a pair of elastic wristbands on each arm for 7 days. Each wristband has a flat button pressing the P6 acupoint, located on the anterior surface of the forearm, approximately three-finger width up from the crease of the wrist between the tendons of the Palmaris longus and flexor carpi radialis.
* Arm III (control group): Patients receive standard antiemetics as in arm I. Patients are assessed periodically by questionnaires.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any cancer

  * Scheduled to receive their first chemotherapy course
  * Scheduled to receive highly, moderately, or low-emetogenic chemotherapy
  * Scheduled to receive a chemotherapy regimen given as a single administration at the beginning of the course repeated in 3-week courses
* Currently receiving adjuvant chemotherapy as outpatient
* Acupressure wristband-naïve (in terms of never having tried such a wristband; may have seen or heard about such wristbands)

PATIENT CHARACTERISTICS:

* Able to perform self care (i.e., no inability to use wristbands appropriately or mental incapacity preventing continuous and optimal use of wristbands) as judged by the investigators
* No liver disease
* No metabolic risk factors for nausea (i.e., electrolyte imbalances causing nausea/vomiting)
* No mechanical risk factors for nausea (i.e., intestinal obstruction)
* No nausea and/or vomiting due to use of opioids
* No lymphedematous arms
* No chronic alcohol use

PRIOR CONCURRENT THERAPY:

* No concurrent radiotherapy
* No concurrent chemotherapy regimens as inpatients

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 699 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of nausea as assessed by the Rhodes Index of Nausea & Vomiting before and after chemotherapy

SECONDARY OUTCOMES:
Incidence and extent of acute and delayed nausea and vomiting by the MASCC Antiemesis Tool at day 10 of each course
Quality of life as assessed by FACT-G at baseline and at day 10 of each course
Anxiety as assessed by the Hospital Anxiety & Depression Scale at baseline
Expectation for nausea and vomiting as assessed by the Patient Expectations of Nausea/Vomiting after each chemotherapy course
Measure of blindness (to intervention vs sham) assessed after chemotherapy
Sociodemographic and treatment characteristics assessed at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molassiotis, MD, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, England, United Kingdom